CLINICAL TRIAL: NCT06286566
Title: Comparison of Osstem TS3 With SOI Surface in Patients With and Without Type 2 Diabetes: A Multicenter Prospective Cohort Study
Brief Title: Soi TS3 Surface in Patients With and Without Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea M. I. Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Assistent Professor, Università degli Studi di Sassari
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_2
Record Dates: First submitted 2023-04-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant; Dental Implant-Abutment Design
Keywords: Dental Implant; Diabetics Patients; SOI Surface

STUDY DESIGN:
Intervention Model Description: Multicenter prospective cohort study
Who Masked: Outcomes Assessor
Masking Description: centralized radiographic assessor, outcome assessors(when possible), and the statistical advisors will be blind to the used implants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetics group (Experimental): Group of subjects with diabetes who will be inserted implants with a new implant surface called SOI
  Interventions: Device: Implant placement with soi surface in diabetic subjects
- Healthy Group (Active Comparator): Group of helthy subjects who will be inserted implants with a new implant surface called SOI to compare them with the group of diabetic subjects
  Interventions: Device: Implant placement with soi surface in healthy subjects

INTERVENTIONS:
Device: Implant placement with soi surface in diabetic subjects — Implants placement with SOI surface in subjects with diabetes who have lost at least one tooth element and need of a prosthetic implant-supported rehabilitation. After osseointegration implants will receive definitive prosthesis.
  Arms: Diabetics group
Device: Implant placement with soi surface in healthy subjects — Implants placement with SOI surface in subjects without diabetes who have lost at least one tooth element and need of a prosthetic implant-supported rehabilitation. After osseointegration implants will receive definitive prosthesis.
  Arms: Healthy Group

SUMMARY:
The aim of this prospective cohort study is to compare clinical and radiographic data of Osstem implants with SOI surface placed in patients with or without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old able to sign an informed consent.
* Patients with at least a single tooth loss in the maxilla or mandible. Patient will provide only one site for the research. Implant sites must allow the placement of implants of at least 3.5 mm (upper laterals and lower incisors); 4 mm (central incisors, canines, and premolars) or 4.5 (molars) mm of diameter and at least 7 mm of length.
* Smokers will be included and categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day).
* Patients with a plaque index (PI) of less than, or equal to 25% at the time of surgery.
* In case of post-extractive sites, they must have been healing for at least 3 months before being treated in the study.
* Only in the test group, patients with controlled type 2 diabetes mellitus with at least 2 years of disease evaluation of HbA1C values between 6% and 10 % at the time of implant placement will be included.
* Only in the control group, healthy patients without any sign of type 2 diabetes mellitus will be included

Exclusion Criteria:

* General contraindications to implant surgery (except for type two diabetes in test group).
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients (except for type two diabetes in test group).
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Previous guided bone reconstruction at the intended implant sites.
* Uncontrolled diabetes (except for type two diabetes in test group).
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of prosthesis failure: | Up to 5 years
  whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reason
Number of implant failure | Up to 5 years
  defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable.
Number of complication | Up to 5 years
  Technical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, suppuration, peri-implantitis, etc.) complication will be considered

SECONDARY OUTCOMES:
Rate of peri-implant marginal bone level changes | At 1,3 and 5 years
  eri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured
Valuation of patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  Would you undergo the same therapy again? Possible answers: "yes" or "no

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tallarico, Rome, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No